CLINICAL TRIAL: NCT05305053
Title: Practice Variation in Preoperative Multidisciplinary Team Discussions for High-risk Noncardiac Surgical Patients in the Netherlands: A Multicenter Prospective Observational Study.
Brief Title: Practice Variation in Preoperative Multidisciplinary Team Discussions
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Jacqueline Vernooij, Principal investigator, Rijnstate Hospital
Other Study IDs: 2021-1952
Record Dates: First submitted 2022-01-18; First posted 2022-03-31 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Pre-operative; High-risk Patient; Frailty
Keywords: high-risk;; preoperative risk prediction; perioperative mortality; Multidisciplinary Team meeting
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high-risk noncardiac surgery patients for preoperative Multidisciplinary Team (MDT) discussion: observation of MDT in 11 hospitals
  Interventions: Other: preoperative MDT discussion

INTERVENTIONS:
Other: preoperative MDT discussion — high-risk patients are subjected to an MDT discussion among care providers

SUMMARY:
Preoperative multidisciplinary team (MDT)discussions are recommended by national and international guidelines. However, no guidance is given on how to organise and execute an MDT discussion. The objective of this study is to describe the methods used for preoperative MDT discussion executed in the Netherlands.

DETAILED DESCRIPTION:
Due to the increase in life expectancy and improved care for patients suffering from a chronic disease, the number of complex patients requiring surgery increases. Surgical treatment is often the optimal treatment to improve survival, but it is important for high-risk patients, to balance the potential benefits of treatment against the risk of potential permanent loss of functional capacity and quality of life. Multidisciplinary Team (MDT) meetings may be a sophisticated solution to discuss the harm-benefit ratio between different caregivers. There are currently no randomized studies comparing preoperative MDT meetings for high-risk non-cardiac surgery patients with no preoperative MDTs. In observational studies, the preoperative MDT altered medical treatment and management in more than 80% of patients, including 13-36% of patients who, after MDT, did not undergo the planned surgical procedure.(1, 2) The implementation of a preoperative MDT for frail patients scheduled for colorectal surgery was associated with a statistically nonsignificant reduction in severe postoperative complications from 33% to 22% of patients or up to 25% changes in care management.(1, 3) In a retrospective study Sroka found that for 36% of the discussed, high-risk cancer patients the case was risk prohibitive. The retrospective study by Vernooij et al. showed that only 27% of discussed patients received care as planned.(4) In cancer care, extensive experience exists with MDT meetings also known as tumor boards. The introduction of MDTs has impacted patient treatment in oncology. However, these tumor boards may be hindered by an excessive caseload and time pressure(5) which may limit a positive effect of MDT meetings on patient outcome.(6) A preoperative MDT may therefore complement these tumor boards since only the high-risk cases are selected for discussion and medical consultants are invited based specifically on the patients' comorbidities.

Several international guidelines have recommended MDT discussions for high-risk patients but they are not widely implemented yet. (7-9) Not executing preoperative MDT meetings may be a consequence of the fact that objective evidence for the value of the preoperative MDT meetings for high-risk, noncardiac patients is practically nonexistent. Also, no guidance exists on how best to organize an MDT meeting. Sroka proposes a protocol for the identification and multidisciplinary discussion of predefined high-risk patients.(2) In the current multicenter observational study in the Netherlands, the aim is to document how preoperative MDT meetings for high-risk non-cardiac surgery patients are executed. For the hospitals where MDT meetings are executed, considerable practice variation between hospitals may exist concerning performing and organizing MDT meetings. The practice variation may exist regarding patient selection, MDT meeting organization and attendance, MDT discussions, decisions made and, lastly, regarding nonsurgical management.

The first objective of this study is to describe the practice variation in executing preoperative MDT meetings in the presence of an anesthesiologist. The research question is: How much and what kind of variation exists in execution of preoperative MDT meetings for high-risk non-cardiac surgical patients. Secondary objectives are: what is the frequency of care management changes ordered by an MDT discussion; how do these changes affect outcome of the patients measured by the frequency of Serious adverse events; 30 day, 3 months and 12 months mortality postoperatively or post MDT discussion; calculated risks; differences in high-risk patient identification and the relation between calculated risks and outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients selected for a Multidisciplinary Team discussion

Exclusion Criteria:

* No implicit consent given for scientific research

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All high risk noncardiac surgical patients selected for a preoperative MDT discussion.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Attendance of the MDT | 1-4-2022 untill 1-10-2022
  number of carers present at meeting
Decisions made in MDT | 01-04-2022 untill 01-010-2022
  number of decisions made
12 months postoperative mortality or post MDT | 01-04-2022 untill 01-10-2024
  number of patients that died within 12 months postoperative or 12 months post MDT

SECONDARY OUTCOMES:
30 day postoperative mortality or post MDT | 01-04-2022 untill 01-10-2022
  number of patients that died within 30 days
Serious adverse events at 12 months postoperative or post MDT | 01-04-2022 untill 01-10-2024
  number of serious adverse events per patient at 12 months postoperative or 12 months post MDT classified by the Clavien Dindo Classification
Hospital admissions at 12 months postoperative or post MDT | 01-04-2022 untill 01-10-2024
  number of hospital admissions per patient at 12 months postoperative or 12 months post MDT

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Vernooij, MD, Principal Investigator — Rijnstate
Locations (9):
- Netherlands (9):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Gelderse Vallei, Ede, Gelderland
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - MC Leeuwarden, Leeuwarden, Provincie Friesland
  - Amsterdam University Medical Centre location VU, Amsterdam, South Holland
  - LUMC, Leiden, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Franciscus Gasthuis, Rotterdam, South Holland
  - UMCU, Utrecht